CLINICAL TRIAL: NCT02805712
Title: Pilot Study of a Focused Palliative Care Intervention for Recently Hospitalized High-Risk Patients With Heart Failure
Brief Title: Focused Palliative Care Intervention in Advanced Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Akshay Desai, MD, Director, Heart Failure Disease Management Program, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2014P001391
Record Dates: First submitted 2016-05-20; First posted 2016-06-20 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Heart Failure; Quality of Life
Keywords: Heart Failure; Palliative Care
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (Active Comparator): Participant will receive usual care for Heart Failure patients, which include standard written material on Advanced Care planning and supportive cardiology/palliative care consult if ordered by attending.
  Interventions: Other: Control
- Verbal Information and Discussion (Experimental): Participants will participate in a guided goals of care conversation and the support of a Palliative Care Social Worker who is working closely with the patients' primary cardiology team. Social worker has ongoing clinical review of participants with a Palliative Care physician who will provide a full medical consult if appropriate.
  Interventions: Other: Verbal Information and Discussion

INTERVENTIONS:
Other: Verbal Information and Discussion — Intervention patient will receive a outpatient session with a palliative care social worker in the heart failure clinic two weeks post discharge consent focusing on goals of care.
  Arms: Verbal Information and Discussion
Other: Control — The control group will receive usual written care material and a palliative care consult if ordered by physician.
  Arms: Control

SUMMARY:
This small pilot study will be assessing the the impact of a standardized, social-worker led, longitudinal palliative care intervention on alignment of patient and physician understanding of prognosis and goals of care. Secondary objectives include assessing the impact of this intervention on documentation of advanced care planning and end of life preferences, symptom burden, quality of life and health care utilization.

DETAILED DESCRIPTION:
Patients will be assigned to one of two groups a) longitudinal goals of care discussion led by a palliative care-trained social worker or b) usual care + written information regarding advanced directives. The intervention group will be enrolled in the hospital and then be followed longitudinally for 3 months by a palliative care-trained social worker who will shepherd a conversation around prognosis, expectations, and goals of care. The results of these conversations will be documented in the electronic medical record and shared with the clinical team. Clinical symptoms that are identified during these conversations will be evaluated by a Palliative Care Physician who will relay suggestions regarding management to the primary treating clinician. Baseline surveys will assess prognostic awareness, symptom burden, anxiety, depression, and quality of life for both groups. At the conclusion of the study, an individualized follow-up plan will be devised for each patient based on a needs assessment by the study social worker.

Patients assigned to the control/usual care arm will complete the same series of questionnaires as those assigned to the intervention group and will undergo usual in hospital and post-discharge treatment as directed by their care team. All control subjects will receive written Advanced Care planning and Heart Failure education materials as provided routinely to inpatients at Brigham and Women's Hospital. At the 6 month visit following hospitalization, these patients will be asked to complete follow up questionnaires and then will be given the option to participate in the above verbal intervention and guided "Goals and Values" conversation that was provided to the intervention group.

ELIGIBILITY:
Inclusion Criteria

* Symptomatic Heart Failure (NYHA II-IV)
* Hospitalized or recently for acute decompensation with at least one of the following high-risk features

  * Prior hospitalization for Heart Failure (HF) within 1 year
  * Age > 80 years
  * Chronic Kidney Disease (estimated Glomerular Filtration Rate (eGFR) < 45 mL/min/m2)
  * Systolic Blood Pressure < 100 mm Hg
  * Serum sodium < 130 meq/L
  * Cardiogenic Shock (Cardiac Index < 2.0)
  * Serious Non-Cardiovascular Illness (e.g. advanced stage cancer, Chronic Obstructive Pulmonary Disease (COPD) , or the like.
* Ability to Provide Informed Consent
* Permission of attending physician

Exclusion Criteria

* Anticipated major cardiac surgery, including Ventricular Assist Device (VAD) or transplant, within 3 months of enrollment
* Already enrolled in hospice or receiving outpatient palliative care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-09; Primary Completion 2016-06 (Actual); Study Completion 2016-12-01 (Actual)

PRIMARY OUTCOMES:
Is there a change in patient understanding of prognosis with the addition of a palliative care intervention? | 6 months
  Assessment tool: Patient Preferences Questionnaire.

SECONDARY OUTCOMES:
Is there an impact on documentation of advanced care planning documentation with a palliative care intervention? | 6 months
  Chart review of Advanced Care Planning documents and written notes by members of clinical team.
Is there an impact on symptom burden through a palliative care intervention? | Three months
  Assessment tool: : The Kansas City Cardiomyopathy Questionnaire (KCCQ-12)
Is there an impact on perceived level of illness through a palliative care intervention? | 6 months
  Assessment tool: EQ visual analogue scale (EQ-VAS)
Is there an impact on overall patient well being through a palliative care intervention? | Three months
  Assessment tool: The Functional Assessment of Chronic Illness Therapy ( FACIT-Sp)
Is there an impact on depression through a palliative care intervention? | 6 months
  Assessment tool: Patient Health Questionnaire (PHQ-8)
Is there an impact on anxiety through a palliative care intervention? | 6 months
  Assessment tool: General Anxiety Disorder (GAD-7)
Is there an impact on cost of treatment through a palliative care intervention? | 6 months
  Focus will be on cost through health care utilization as aggregated by number of hospital days, days in ICU and 30 day re-admissions.

CONTACTS AND LOCATIONS:
Overall Officials: Akshay S Desai, MPH, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] O'Donnell AE, Schaefer KG, Stevenson LW, DeVoe K, Walsh K, Mehra MR, Desai AS. Social Worker-Aided Palliative Care Intervention in High-risk Patients With Heart Failure (SWAP-HF): A Pilot Randomized Clinical Trial. JAMA Cardiol. 2018 Jun 1;3(6):516-519. doi: 10.1001/jamacardio.2018.0589. PMID 29641819